CLINICAL TRIAL: NCT03273712
Title: Phase II, Dosimetry Guided, Peptide Receptor Radiotherapy (PRRT) Using 90Y-DOTA tyr3-Octreotide (90Y-DOTATOC) in Children and Adults With Neuroendocrine and Other Somatostatin Receptor Positive Tumors
Brief Title: Dosimetry-Guided, Peptide Receptor Radiotherapy (PRRT) With 90Y-DOTA- tyr3-Octreotide (90Y-DOTATOC)
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of Iowa (Other)
Collaborators: National Institutes of Health (NIH) (NIH); National Cancer Institute (NCI) (NIH)
Responsible Party: Principal Investigator, Sue O'Dorisio, Professor, University of Iowa
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 201708778; R01CA167632 (NIH); 201412770 (Other: University of Iowa); NCT02441088 (obsolete NCT alias)
Record Dates: First submitted 2017-09-01; First posted 2017-09-06 (Actual); Results first posted 2023-02-09 (Actual); Last update posted 2023-02-09 (Actual); Status verified 2023-02

CONDITIONS: Neuroendocrine Tumors; Meningioma; Neuroblastoma; Medulloblastoma
MeSH Terms: conditions — Neuroendocrine Tumors; Meningioma; Neuroblastoma; Medulloblastoma | interventions — 90Y-octreotide, DOTA-Tyr(3)-; Whole Body Imaging; Amino Acids; arginyllysine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- 90Y-DOTA-tyr3-Octreotide (Experimental): Patients will receive 3 doses of 90YDOTATOC followed by 90Y-DOTATOC PET scans, with 6 -8 weeks between doses. They will be followed for 6-9 months after the last treatment dose. CT or MRI scans will be given at the 3 month and 6-9 month followups plus a 68Ga-DOTATOC or DOTATATE PET scan at the 6-9 month followup. The exact dose of 90YDOTATOC therapy for each patient will be determined by dosimetry.
  Interventions: Radiation: 90Y-DOTA tyr3-Octreotide; Diagnostic Test: 68Ga-DOTATOC PET Positron Emission Tomography (PET) whole body scan; Drug: Amino Acids

INTERVENTIONS:
Radiation: 90Y-DOTA tyr3-Octreotide — 90Y-DOTATOC is a radiopharmaceutical that will be used as a treatment for both children and adults with neuroendrocrine and other somatostatin receptor positive tumors.
  Other Names: 90Y-DOTATOC
Diagnostic Test: 68Ga-DOTATOC PET Positron Emission Tomography (PET) whole body scan — 68Ga-DOTATOC is a radiopharmaceutical used in PET scans to identify tumors as it can adhere to Somatostatin Receptors.
Drug: Amino Acids — This is a solution of amino acids that will decrease the amount of 90Y-DOTATOC that recirculates through the body after injection, therefore decreasing the radiation dose to the kidneys.
  Other Names: Lysine and Arginine

SUMMARY:
This is a Phase 2 peptide receptor radionuclide therapy trial of 90Y-DOTATOC in patients with somatostatin receptor positive tumors.

DETAILED DESCRIPTION:
This is a Phase 2 peptide receptor radionuclide therapy trial of 90Y-DOTATOC in patients with somatostatin receptor positive tumors. The somatostatin receptor targeting of the therapeutic will be checked with 68Ga-DOTATOC PET-CT imaging prior to therapy. Treatment consists of 3 cycles, 6-8 weeks apart. Cycle 1 dose is fixed with Cycles 2 and 3 doses to be determined by dosimetry-based calculation of renal doses from previous cycles not to exceed 23 Gy for the total renal dose.

The goals of this project are to

1. Demonstrate the safety and efficacy of dosimetry-guided peptide receptor radiotherapy using 90Y-DOTA-tyr3-Octreotide in patients with neuroendocrine and other somatostatin receptor expressing tumors.
2. Monitor all adverse events associated with peptide receptor radiotherapy using 90Y-DOTATOC.
3. Establish 68Ga-DOTA-tyr3-Octreotide (68Ga-DOTATOC) or 68Ga-DOTATATE PET/CT as an accurate technique for diagnosis, staging, treatment targeting, and monitoring response to 90Y-DOTATOC therapy.

ELIGIBILITY:
Inclusion Criteria:

1. Disease not amenable to standard treatment (nonresectable or disease present after one or more surgeries and/or Sandostatin treatment) or subject has failed existing first line chemotherapy, biologic therapy, targeted agent therapy or radiation therapy.
2. Participation in Iowa Neuroendocrine Tumor Registry.
3. A pathologically confirmed (histology or cytology) malignant neoplasm with at least one target lesion that is confirmed by conventional imaging and is determined to express somatostatin receptors by 68Ga-DOTATOC (TATE) PET within 6 months prior to treatment with 90Y-DOTATOC.
4. The target lesion is one that either has never received external beam radiation or has been previously irradiated and has since demonstrated progression. Any local irradiation of the target lesion or any non-target lesions via external beam, conformal or stereotactic radiation treatments must have occurred more than 4 weeks prior to study drug administration. Any full cranial-spinal radiation, whether or not a target lesion is included in the field, must have occurred more than 3 months prior to study drug administration.
5. Life expectancy > 2 months at the time of study drug administration.
6. Archival tissue from a previous biopsy will be required.
7. Age ≥ 6 months-90 years at the time of study drug administration.
8. Performance status as determined by Karnofsky ≥ 60 or Lansky Play Scale ≥ 60% at the time of study drug administration.
9. Completion of Norfolk Quality of Life Questionnaire.
10. Within 7-10 days of study drug administration, patients must have normal organ and marrow function as defined below:

    * absolute neutrophil count >1000/mm3
    * Platelets >90,000/mm3
    * total bilirubin <3X ULN for age
    * AST(SGOT) & ALT(SGPT) <10X institutional upper limit of normal for age
    * Urinalysis no greater than 1+ hematuria or proteinuria
    * Renal function* Adults(age18 or >): Serum creatinine ≤ 1.2 mg/dl; if serum creatinine is >1.2 mg/dL, nuclear GFR will be measured. GFR will need to be ≥ 80 ml/min/1.73m2 for subjects ≤40 years old, ≥ 70 ml/min/1.73m2 for subjects between 41-50; ≥ 60 ml/min/1.73m2 for subjects between 51-60; ≥ 50 ml/min/1.73m2 for subjects > 60 years old.

    Children(age <18): nuclear GFR ≥ 80 mL/min/1.73 m2

    * Renal function criteria based on our previous experience with 90Y-DOTATOC therapy and known changes in GFR with age13,21,33-35
11. The effects of 90Y-DOTA-tyr3-Octreotide on the developing human fetus are unknown. For this reason and because Class C agents are known to be teratogenic, women and men of child-bearing potential must agree to use adequate contraception (hormonal or barrier method of birth control) prior to study entry and for the duration of study participation. Should a woman become pregnant or suspect she is pregnant while participating in this study, she should inform her treating physician immediately.
12. Ability to understand and the willingness to sign a written informed consent document.

Exclusion Criteria:

1. Pregnant women are excluded from this study because 90Y-DOTATOC is a Class C agent with potential teratogenic or abortifacient effects.
2. Because there is an unknown but potential risk for adverse events in nursing infants secondary to treatment of the mother with 90Y-DOTATOC, breastfeeding should be discontinued until 6 weeks after the last administration of study drug.
3. Surgery within 4 weeks of study drug administration.
4. External beam radiation to both kidneys (scatter doses of <500 cGy to a single kidney or radiation to < 50% of a single kidney is acceptable).
5. Prior PRRT with 90Y-DOTATOC (TATE) or 177Lu-DOTATOC (TATE) or 131I-MIBG therapy for this malignancy.
6. Another investigational drug within 4 weeks of study drug administration.
7. Concurrent, malignant disease for which patient is on active therapy.
8. Another significant medical, psychiatric, or surgical condition which is currently uncontrolled by treatment and which would likely affect the subject's ability to complete this protocol.
9. Any subject for whom, in the opinion of their physician, a 12-hour discontinuation of somatostatin analogue therapy represents a health risk. Also subjects who have received SandostatinLAR in the past 28 days or long-acting lanreotide within the past 8 weeks are excluded. Subjects may be maintained on short acting octreotide during the time from last injection of long-acting somatostatin analogue until 12 hrs prior to injection of study drug. Known antibodies to Octreotide, Lanreotide, or DOTATOC or history of allergic reactions attributed to compounds of similar chemical or biologic composition to 90Y-DOTATOC.
10. Patients who have had chemotherapy within 4 weeks (6 weeks for nitrosoureas or mitomycin C) of study drug administration or those who have not recovered from adverse events due to agents administered more than 4 weeks earlier.
11. Uncontrolled illness including, but not limited to ongoing or active infection, symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia, or psychiatric illness/social situations that would limit compliance with study requirements.
12. Subject weighs more than 450 pounds. (Subjects who weigh more than 450 pounds will not be able to fit inside the imaging machines.)
13. Inability to lie still for the entire imaging time (due to cough, severe arthritis, etc.)

Ages: 6 Months to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 39 (Actual)
Dates: Start 2017-09-29 (Actual); Primary Completion 2020-05-27 (Actual); Study Completion 2020-05-27 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: M. Sue O'Dorisio, MD, PhD, Principal Investigator — University of Iowa
Locations (1):
- University of Iowa Hospitals and Clinics, Iowa City, Iowa, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The University of Iowa Neuroendocrine Tumor Registry includes over 1500 individuals with NETs who have signed consent to be contacted when new clinical trials are available. The University of Iowa Children's Hospital has children with neuroblastoma and medulloblastoma (or other brain tumor) and neuroendocrine tumor who may be interested; in this case, participation would be offered only if/when the child failed conventional therapy.
Pre-assignment Details: A subject can have the 90Y-DOTATOC treatment the next day after he/she signs the consent. Administration of 90Y-DOTATOC will likely be 12 hours to 1 month following confirmation of positive lesions on 68Ga-DOTATOC PET scan.
Period: Overall Study
Arm/Group | 90Y-DOTA-tyr3-Octreotide
Started | 39
Completed | 32
Not Completed | 7
Not completed — Death | 5
Not completed — Adverse Event | 1
Not completed — Disease Progression | 1

BASELINE CHARACTERISTICS:
Arm/Group | 90Y-DOTA-tyr3-Octreotide
Number analyzed (Participants) | 39
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 4
  Between 18 and 65 years | 24
  >=65 years | 11
Age, Continuous [Mean (Full Range); unit: years] | 54 [9 to 79]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 19
  Male | 20
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 39
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 2
  White | 37
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 39

OUTCOME MEASURES:

1. Primary Outcome: Frequency of Tumor Response at 9 Months After Last Treatment
Description: Response Evaluation Criteria In Solid Tumors Criteria (RECIST v1.1) was used to quantify tumor response by comparison of baseline and last follow-up visit (6-9 months after last treatment) diagnostic CT/MRI scans.
Time Frame: Baseline through last follow-up visit (6-9 months after last treatment), up to approximately 10-13 months.
Measure: Count of Participants; unit: Participants
Arm/Group | 90Y-DOTA-tyr3-Octreotide
Number analyzed (Participants) | 39
Participants
  Complete Response | 0
  Partial Response | 1
  Stable Disease | 19
  Progressive Disease | 15
  Not Evaluable | 4

2. Primary Outcome: Percentage of Patients With Grade 4 or Higher Renal Adverse Event.
Description: The percentage of patients who experience a grade 4 or higher renal adverse event. Renal adverse events were graded using CTCAE v4.0 criteria.
Time Frame: Initiation of treatment through last follow-up visit (6-9 months after last treatment), up to approximately 10-13 months.
Measure: Count of Participants; unit: Participants
Arm/Group | 90Y-DOTA-tyr3-Octreotide
Number analyzed (Participants) | 39
Participants | 0

3. Primary Outcome: Percentage of Patients With Grade 4 or Higher Irreversible Adverse Events
Description: The percentage of patients who experience a grade 4 or higher irreversible adverse event. Adverse events were graded using CTCAE v4.0 criteria.
Time Frame: as for outcome 2
Measure: Count of Participants; unit: Participants
Groups:
- 90Y-DOTA-tyr3-Octreotide: Patients will receive 3 doses of 90YDOTATOC, with 6 -8 weeks between doses. They will be followed for 6 monthsafter the last treatment dose. CT or MRI scans will be given at the 3 month and 6 month followups. The exact dose of 90YDOTATOC therapy for each patient will be determined by dosimetry.
  90Y-DOTA tyr3-Octreotide: 90Y-DOTATOC is a radiopharmaceutical that will be used as a treatment for both children and adults with neuroendrocrine and other somatostatin receptor positive tumors.
  Amino Acids: This is a solution of amino acids that will decrease the amount of 90Y-DOTATOC that recirculates through the body after injection, therefore decreasing the radiation dose to the kidneys.
Arm/Group | 90Y-DOTA-tyr3-Octreotide
Number analyzed (Participants) | 39
Participants | 0

ADVERSE EVENTS:
Time Frame: Adverse even documentation began after radiotracer injection and continues through 1 calendar day following imaging, up to approximately 10-13 months
Arm/Group | 90Y-DOTA-tyr3-Octreotide
All-Cause Mortality (participants affected / at risk) | 5/39
Serious Adverse Events (participants affected / at risk) | 14/39
Other Adverse Events (participants affected / at risk) | 37/39
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | 90Y-DOTA-tyr3-Octreotide (N=39)
Anemia (Blood and lymphatic system disorders) | 1 (2)
Atrioventricular block complete (Cardiac disorders) | 1 (1)
Endocrine disorders - Other, specify (Endocrine disorders) | 1 (2)
Nausea (Gastrointestinal disorders) | 1 (1)
Small intestinal obstruction (Gastrointestinal disorders) | 2 (3)
Edema limbs (General disorders) | 1 (3)
Pain (General disorders) | 1 (1)
Bronchial infection (Infections and infestations) | 1 (1)
Catheter related infection (Infections and infestations) | 1 (1)
Infections and infestations - Other, specify (Infections and infestations) | 1 (2)
Sepsis (Infections and infestations) | 2 (2)
Urinary tract infection (Infections and infestations) | 1 (1)
Fall (Injury, poisoning and procedural complications) | 1 (1)
Alanine aminotransferase increased (Investigations) | 1 (3)
Aspartate aminotransferase increased (Investigations) | 1 (3)
Blood bilirubin increased (Investigations) | 1 (3)
Creatinine increased (Investigations) | 1 (1)
Platelet count decreased (Investigations) | 1 (3)
Hyperglycemia (Metabolism and nutrition disorders) | 1 (1)
Hyperkalemia (Metabolism and nutrition disorders) | 1 (1)
Hypokalemia (Metabolism and nutrition disorders) | 1 (1)
Musculoskeletal and connective tissue disorder - Other, specify (Musculoskeletal and connective tissue disorders) | 1 (1)
Neoplasms benign, malignant and unspecified (incl cysts and polyps) - Other, specify (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (2)
Dizziness (Nervous system disorders) | 1 (2)
Headache (Nervous system disorders) | 1 (1)
Syncope (Nervous system disorders) | 1 (1)
Renal and urinary disorders - Other, specify (Renal and urinary disorders) | 1 (1)
Vascular disorders - Other, specify (Vascular disorders) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | 90Y-DOTA-tyr3-Octreotide (N=39)
Anemia (Blood and lymphatic system disorders) | 7 (7)
Atrioventricular block complete (Cardiac disorders) | 1 (1)
Cardiac disorders - Other, specify (Cardiac disorders) | 1 (1)
Ear and labyrinth disorders - Other, specify (Ear and labyrinth disorders) | 1 (1)
Endocrine disorders - Other, specify (Endocrine disorders) | 4 (5)
Eye disorders - Other, specify (Eye disorders) | 2 (2)
Abdominal distension (Gastrointestinal disorders) | 1 (1)
Abdominal pain (Gastrointestinal disorders) | 9 (12)
Constipation (Gastrointestinal disorders) | 2 (2)
Diarrhea (Gastrointestinal disorders) | 3 (4)
Gastritis (Gastrointestinal disorders) | 1 (1)
Gastrointestinal disorders - Other, specify (Gastrointestinal disorders) | 1 (1)
Gastroparesis (Gastrointestinal disorders) | 1 (2)
Hemorrhoidal hemorrhage (Gastrointestinal disorders) | 1 (1)
Nausea (Gastrointestinal disorders) | 37 (83)
Oral dysesthesia (Gastrointestinal disorders) | 1 (1)
Small intestinal obstruction (Gastrointestinal disorders) | 2 (2)
Upper gastrointestinal hemorrhage (Gastrointestinal disorders) | 1 (1)
Vomiting (Gastrointestinal disorders) | 15 (26)
Chills (General disorders) | 3 (3)
Edema face (General disorders) | 1 (1)
Edema limbs (General disorders) | 1 (1)
Fatigue (General disorders) | 15 (20)
Fever (General disorders) | 5 (5)
Flu like symptoms (General disorders) | 1 (1)
Gait disturbance (General disorders) | 1 (1)
General disorders and administration site conditions - Other, specify (General disorders) | 1 (1)
Infusion site extravasation (General disorders) | 5 (6)
Injection site reaction (General disorders) | 1 (1)
Localized edema (General disorders) | 1 (1)
Non-cardiac chest pain (General disorders) | 1 (1)
Pain (General disorders) | 2 (2)
Hepatobiliary disorders - Other, specify (Hepatobiliary disorders) | 1 (1)
Bronchial infection (Infections and infestations) | 2 (2)
Catheter related infection (Infections and infestations) | 1 (1)
Infections and infestations - Other, specify (Infections and infestations) | 2 (3)
Sepsis (Infections and infestations) | 2 (2)
Skin infection (Infections and infestations) | 1 (1)
Urinary tract infection (Infections and infestations) | 1 (1)
Fall (Injury, poisoning and procedural complications) | 1 (1)
Alanine aminotransferase increased (Investigations) | 1 (2)
Blood bilirubin increased (Investigations) | 1 (2)
Creatinine increased (Investigations) | 1 (1)
Investigations - Other, specify (Investigations) | 1 (1)
Lymphocyte count decreased (Investigations) | 5 (5)
Neutrophil count decreased (Investigations) | 3 (6)
Platelet count decreased (Investigations) | 4 (4)
Weight gain (Investigations) | 3 (3)
White blood cell decreased (Investigations) | 4 (8)
Dehydration (Metabolism and nutrition disorders) | 2 (3)
Hyperglycemia (Metabolism and nutrition disorders) | 1 (1)
Hyperkalemia (Metabolism and nutrition disorders) | 2 (3)
Arthralgia (Musculoskeletal and connective tissue disorders) | 3 (3)
Back pain (Musculoskeletal and connective tissue disorders) | 2 (3)
Bone pain (Musculoskeletal and connective tissue disorders) | 1 (1)
Flank pain (Musculoskeletal and connective tissue disorders) | 1 (1)
Musculoskeletal and connective tissue disorder - Other, specify (Musculoskeletal and connective tissue disorders) | 1 (1)
Myalgia (Musculoskeletal and connective tissue disorders) | 2 (2)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 2 (2)
Neoplasms benign, malignant and unspecified (incl cysts and polyps) - Other, specify (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (2)
Dizziness (Nervous system disorders) | 6 (9)
Headache (Nervous system disorders) | 8 (10)
Lethargy (Nervous system disorders) | 1 (1)
Memory impairment (Nervous system disorders) | 1 (1)
Paresthesia (Nervous system disorders) | 1 (1)
Peripheral sensory neuropathy (Nervous system disorders) | 1 (1)
Syncope (Nervous system disorders) | 1 (1)
Anxiety (Psychiatric disorders) | 2 (3)
Insomnia (Psychiatric disorders) | 1 (1)
Renal and urinary disorders - Other, specify (Renal and urinary disorders) | 1 (1)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Flushing (Vascular disorders) | 1 (1)
Hypertension (Vascular disorders) | 3 (4)
Vascular disorders - Other, specify (Vascular disorders) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2019-08-19): https://cdn.clinicaltrials.gov/large-docs/12/NCT03273712/Prot_SAP_000.pdf
  • Informed Consent Form (2019-07-27): https://cdn.clinicaltrials.gov/large-docs/12/NCT03273712/ICF_001.pdf